CLINICAL TRIAL: NCT03051373
Title: Phase 2 Trial of Nab-paclitaxel Plus S-1 vs Gemcitabine Plus Cisplatin as 1-line Chemotherapy of Patients With Local Advanced and/or Metastatic Transitional Cell Carcinoma of Urothelial Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Bo Yang, Associate Chief Doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BY-001
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Carcinoma, Transitional Cell
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Taxes; S 1 (combination); Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nab-paclitaxel plus S-1 (Experimental): Nanoparticle albumin-bound paclitaxel is given at 120mg/m2 intravenously over 30 minutes on day 1 and 8, in combination with S-1 which is orally administered (40-60 mg according to the body surface, Bid) on day 1-14 of each 21-days cycle. Number of cycle: 6 cycles.
  Interventions: Drug: nanoparticle albumin-bound paclitaxel, S-1
- Gemcitabine plus cisplatin (Active Comparator): Gemcitabine is given at 1000mg/m2 combination with cisplatin 75mg/m2 intravenously on day 1 and 8 of each 21-days cycle. Number of cycle: 6 cycles.
  Interventions: Drug: Gemcitabine, cisplatin

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel, S-1 — Nanoparticle albumin-bound paclitaxel is given at 120mg/m2 intravenously over 30 minutes on day 1 and 8, in combination with S-1 which is orally administered (40-60 mg according to the body surface, Bid) on day 1-14 of each 21-days cycle. Number of cycle: 6 cycles.
  Other Names: nab-paclitaxel abraxane ABI-007
  Arms: nab-paclitaxel plus S-1
Drug: Gemcitabine, cisplatin — Gemcitabine is given at 1000mg/m2 combination with cisplatin 75mg/m2 intravenously on day 1 and 8 of each 21-days cycle. Number of cycle: 6 cycles.
  Other Names: GEMXAR
  Arms: Gemcitabine plus cisplatin

SUMMARY:
Gemcitabine plus cisplatin have been the most studied and used anticancer agents in patients with local advanced and/or metastatic transitional cell carcinoma of urothelial tract even if clinical benefits and survival remains limited.

The purpose of this study is to test in a randomized trial enrolling patients for comparing the efficacy and safety of nab-paclitaxel plus S-1 with Gemcitabine plus cisplatin, in order to determine the most promising agents as the first line treatment of advanced and/or metastatic transitional cell carcinoma of urothelial tract.

DETAILED DESCRIPTION:
Gemcitabine plus cisplatin have been the most studied and used anticancer agents in patients with local advanced and/or metastatic transitional cell carcinoma of urothelial tract even if clinical benefits and survival remains limited.

The purpose of this study is to test in a randomized trial enrolling patients for comparing the efficacy and safety of nab-paclitaxel plus S-1 with Gemcitabine plus cisplatin, in order to determine the most promising agents as the first line treatment of advanced and/or metastatic transitional cell carcinoma of urothelial tract.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form.
2. Man or woman aged 18 years to 70 years.
3. Histologically confirmed unresectable locally advanced or metastatic transitional cell carcinoma, occur in renal pelvis, ureter, urinary bladder or urethra: unresectable stage T3-4 tumor; lymph node metastasis; distance metastasis.
4. Patients with mixed histology may be enrolled if the proportion of transitional cell carcinoma is the predominant component (> 50% of the histopathology sample).
5. Patient without prior anticancer therapy, except for radical excision. Prior adjuvant therapy is allowed, only if the documented relapse intervention >12 months since completion of the last adjuvant therapy.
6. At least one measurable tumor lesion (measurable disease, as defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1), and the measurable tumor received no local therapy (e.g. radiotherapy or cryotherapy).
7. Eastern Cooperative Oncology Group (ECOG) 0-1, no progression within 2 weeks before enter into the trial, and with life expectation of no less than 12 weeks.
8. Patients must have received no previous chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-fluorouracil or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
9. Females of childbearing potential must have a negative serum pregnancy test and must not breast-feed before the first dose. Male also need contraception.

Exclusion Criteria:

1. Patients who accepted any therapy blow:

   * Patients who received prior systemic therapy, including chemotherapy, biotherapy, immunotherapy or experimental therapy, but except for adjuvant and neoadjuvant therapy.
   * Undergo major surgery (except for revascularization) within 4 weeks prior to the first dose.
   * Undergo radiotherapy to more than 30% of marrow, or large field irradiation within 4 weeks prior to the first dose.
   * Patients who were taking (or can't stop within 1 weeks prior to the first dose) any certain drug or herbal supplements, which was known to be the inhibitor or inducer of cytochrome P450 (CYP) 3A4.
   * Other anticancer therapy.
   * The interval from the discontinuation of other investigational agent is less than 5 T1/2 of the drug.
   * Patients were aware of receiving any similar therapy before.
2. Concurrent or past history of another malignancy, need therapy within 2 years after the first dose.
3. Any unresolved AE grade >1 (CTCAE) from previous systemic therapy (e.g. adjuvant chemotherapy) before entry the trial, except for alopecia and grade 2 neuropathy induced by former chemotherapy.
4. Patients with symptomatic central nervous system (CNS) metastasis.
5. Patients with unstable or serious concurrent medical conditions are excluded. The researcher evaluates that the patient who is not suitable for participation in the study. Patients with active infection, but not limited in HBV, HCV, or HIV.
6. Uncontrollable nausea, vomit, chronic gastrointestinal disorders leading to unable to swallow drugs, which may affect the fully absorption of S-1.
7. Patients have active cardiac disease including any of the following:

   * In resting state, average correction QTc > 470 msec on mean value of 3 times screening ECGs, all data come from outpatient screening period.
   * Any clinically significant abnormal ECG form, for example, complete left bundle branch block, 3-degree atrioventricular block, 2-degree atrioventricular block, or PR interval > 250 msec.
   * Any factors may increase the risk of QTc prolongation or arrhythmic event.
8. Marrow function abnormalities and organ dysfunction, reach any of the following laboratory values:

   * ANC <1.5 x 109/L
   * Platelets < 100 x 109/L
   * Hemoglobin < 9.0 g/dL
   * Alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN) without liver metastases; or ALT > 5 x ULN, if liver metastases are present.
   * Aspartate aminotransferase (AST) > 2.5 ULN, without liver metastases; or AST > 5 x ULN, if liver metastases are present.
   * Serum total bilirubin > 1.5 x ULN without liver metastases; or total bilirubin > 3.0 x ULN in patients with well documented Gilbert syndrome or liver metastases.
   * Serum creatinine > 1.5 x ULN with 24-hour clearance < 50 mL/min (measured values, or calculate by the Cockcroft-Gault formula) at the same time; only if creatinine > 1.5 x ULN, 24-hour clearance is needed to be confirmed.
9. Patients who are unwilling or unable to abide by the study protocol, prohibition and requirement. Patient should not take part in the study as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | up to 12 months
  Measure the time of progression-free from start of treatment, assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1

SECONDARY OUTCOMES:
Overall response rate | every 2 cycles (6 weeks) until treatment discontinuation, an expected average of 1 year.
  The proportion of patients with a confirmed complete or partial response (CR or PR) according to RECIST v1.1. CR = disappearance of all target lesions. PR = at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Disease control rate | change from baseline in tumor assessment at 18 weeks (cycle 6).
  Defined by RECIST criteria (version 1.1) as a percentage of best overall responses of CR+PR+SD.
Overall survival | every 8 weeks until disease progression or death on study, an expected average of 2 years. Patients with progressive disease will be followed every 3 months for the first year and every 6 months thereafter up to 5 years.
  Measure of time from Day 1 of study drug administration to disease progression or death or lost to follow-up on study.
The number of treatment-emergent adverse events (AEs) and serous adverse events (SAEs) as a measure of safety | every 3 weeks until treatment discontinuation plus 30 days, an expected average of 1 year.
  The reported incidence of AEs and SAEs with an onset on or after the initiation of therapy will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China